CLINICAL TRIAL: NCT06384443
Title: Inappropriate Use of Proton Pump Inhibitors in Patients With Liver Cirrhosis
Brief Title: Proton Pump Inhibitors in Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: 01001099646
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Proton Pump Inhibitor Adverse Reaction; Liver Cirrhosis
Keywords: Proton pump inhibitors; liver cirrhosis; spontaneous bacterial peritonitis; hepatic encephalopathy; portal hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy; Hypertension, Portal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Inappropriate use of PPI: PPI is prescribed without approved indication or used for a prolonged period beyond the recommended duration.
- Appropriate use of PPI: PPI is prescribed for the approved indication and used within the recommended duration.

SUMMARY:
Proton pump inhibitors (PPIs) inappropriate use, in patients with cirrhosis, presents a significant clinical challenge. This study evaluates overprescription and misuse of PPIs in cirrhotic patients. The patterns of use of PPIs will be classified into two groups based on adherence to the proven indications: Group A: Inappropriate use of PPI, Group B: Appropriate use of PPI. We will estimate the prevalence of PPI misuse in cirrhotics and correlate it with different factors.

DETAILED DESCRIPTION:
The inappropriate use of PPIs in cirrhosis patients is a growing concern. Evidence supporting the use of PPIs in cirrhosis-related conditions is limited. Several adverse outcomes have been linked to PPI use in cirrhosis, including an increased risk of spontaneous bacterial peritonitis and hepatic encephalopathy.

The study aimed to assess the appropriateness of prescribing PPIs to patients with cirrhosis, examining its impact on prescribing practices and identifying associated factors.

in this observational, descriptive, cross-sectional study, cirrhotic patients receiving proton pump inhibitors will be included in the study. Enrolled patients will classified according to the indication for PPI administration: Group A: Inappropriate use of PPI, Group B: Appropriate use of PPI. Use of PPI will be considered inappropriate when prescribed without approved indication or used for a prolonged period beyond the recommended duration. The prevalence of PPI misuse in cirrhotics will be estimated and multivariate analyses will be conducted in order to identify independent predictors of inappropriate use of PPI.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving proton pump inhibitors at the time of enrollment.

Exclusion Criteria:

* Refusal to sign the informed consent form or failure to provide the required information

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a histological, biochemical, imaging and/or clinical data of cirrhosis
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Inappropriate use of PPIs | Six weeks after study completion
  Explore the prevalence of using PPIs without approved indication or for a prolonged period beyond the recommended duration in patients with liver cirrhosis
Predictors for inappropriate use of PPIs | Eight weeks after study completion
  Determine independent predictors of inappropriate use of PPIs in patients with liver cirrhosis using multivariate analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gasser I El-Azab, M.D., Principal Investigator — National Liver Institute, Menoufia University
Locations (1):
- National Liver institute - Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Azab G, Zakareya T, Abdel Aleem M, Edrees A. Inappropriate use of proton pump inhibitors in patients with liver cirrhosis: a cross-sectional study. Eur J Gastroenterol Hepatol. 2025 Oct 1;37(10):1141-1146. doi: 10.1097/MEG.0000000000002985. Epub 2025 Apr 29. PMID 40359285